CLINICAL TRIAL: NCT04449588
Title: A Multi-center, Open-label, Randomized Parallel Controlled Evaluation on the Efficacy and Safety of BDB-001 Injection in the Treatment of Progressive Severe COVID-19 in Phase II/III
Brief Title: Efficacy and Safety Study of BDB-001 in Severe COVID-19 With ALI/ARDS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to the COVID-19 epidemic situation, the sponsor has decided to terminate the project.
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Collaborators: Beijing Defengrui Biotechnology Co. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STS-BDB001-04
Record Dates: First submitted 2020-06-26; First posted 2020-06-29 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; Severe Pneumonia; ALI/ARDS
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — BDB001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Drug: BDB-001 Injection
- Control group (Experimental)
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Drug: BDB-001 Injection — BDB-001 Injection+Conventional treatment
  Arms: Treatment group
Other: Conventional treatment — Conventional treatment only. Local guidelines should be integrated to choose the best supportive care.
  Arms: Control group

SUMMARY:
This multi-center, open, randomized study will evaluate the efficacy and safety of BDB-001 injection in severe COVID-19 with severe pneumonia, or acute lung injury/acute respiratory distress syndrome. Patients will be randomized to two treatment arms (Arm A: Conventional treatment + BDB-001; Arm B: Conventional treatment alone).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 80 years old, both men or women.
2. Confirmed SARS-CoV-2 infection, and meet at least one of the following criteria:

   Confirmed severe COVID-19 in no more than 5 days who meets any of the following criteria:
   1. Respiratory distress, RR ≥ 30 times/min
   2. Finger oxygen saturation (SpO2) ≤93% in resting state(room air)
   3. Arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) ≤ 300 mmHg (1 mmHg = 0.133kpa) in supine position
   4. Pulmonary imaging shows lesion progression > 50% within 24-48 hours.

   Symptoms,signs or chest imaging indicates ALI/ARDS;
3. Requiring a mask oxygen therapy,high-flow nasal cannula oxygen therapy(HFNC).
4. The informed consent form signed.

Exclusion Criteria:

Subject who meets any of the following criteria will be excluded from the trial:

1. Subjects already progressed into critically severe COVID-19 Critical severe standards refer to FDA guidelines,as shown in Appendix 4 or sepsis and sepsis shock.
2. Concomitant with the following situation:severe lung disease such as chronic obstructive pulmonary disease (moderate to severe type), lung cancers, active tuberculosis; severe cardiovascular and cerebrovascular disease: unstable angina pectoris, myocardial infarction, postcardiac surgery, cardiac function ≥ grade 3 (NYHA Classification), or had undergone heart surgery within 6 months before randomization; severe liver diseases (e.g. Child-Pugh score ≥ grade C); severe kidney diseases, such as renal insufficiency (GFR ≤ 15 mL/min/1.73m^2); immune deficiencies or immune-related diseases : including organ or bone marrow transplantation, some autoimmune diseases, IgG4-related diseases, allergic alveolitis, vasculitis; malignancies.
3. Subjects on current treatment with a complement inhibitor such as eculizumab within 1 month before randomization.
4. Subjects with hypersensitivity history to any ingredient contained in the drug.
5. A subject has used the following drugs within 2 weeks prior to screening procedures:

   * Calcineurin inhibitors (e.g., ciclosporin, tacrolimus, etc.)
   * Proliferation inhibitors (e.g., everolimus, sirolimus, etc.)
   * Anti-metabolic drugs (e.g., mycophenolate mofetil, mycophenolate, purine sulphate, etc.)
   * Recombinant human granulocyte macrophage colony stimulating factor (rhGM-CSF)/recombinant human granulocyte colony stimulating factor (rhG-CSF)
6. Pregnant or lactating woman.
7. Subjects who have participated in other interventional clinical trials in the last 3 months or during this trial.
8. Any other circumstances that the investigator considers inappropriate for the participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Time to recovery of peripheral capillary oxygen saturation (SpO2) from baseline | Baseline to Day 28

SECONDARY OUTCOMES:
28-day all-cause mortality rate | Baseline to Day 28
Percentage of patients who progress to critical severe | Baseline to Day 28
Percentage of subjects achieving recovery in SpO2 | Baseline to Day 28
Mean change of PaO2/FiO2 | Baseline to Day 28
Mechanical ventilation time | Baseline to Day 28
Time of oxygen therapy | Baseline to Day 28
Change in inflammation indicators (CRP or IL-6 etc.) from baseline | Baseline to Day 28
Improvement in body temperature | Baseline to Day 28
Mean change from baseline in the clinical improvement based on ordinal scale recommended by the WHO R&D Blueprint during treatment period | Baseline to Day 28
Improvement at D3, 7, 11 & D14 based on ordinal scale recommended by the WHO R&D Blueprint during treatment period | Baseline，Day 3，Day 7，Day 11，Day 14
Time to get categories 1 to 4 in the 8-points ordinal scale | Baseline to Day 28
Time to attain an improvement of 1 point on the ordinal scale | Baseline to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Qing Mao, Ph.D, Principal Investigator — Southwest Hospital of Chongqing
Locations (12):
- Bangladesh (2):
  - Asgar Ali Hospital, Dhaka
  - Bangladesh Specialized Hospital, Dhaka
- Southwest Hospital Chongqing, Chongqing, Chongqing Municipality, China
- India (2):
  - Noble Hospital Pvt Ltd, Nagpur
  - Government Medical College and Hospital, Pune
- Indonesia (3):
  - RSUD Cengkareng(Cengkareng General Hospital), Jakarta, Jakrata
  - RSUD Pasar Minggu(Pasar Minggu General Hospital), Jakarta
  - RSUP Persahabatan(Persahabatan General Hospital), Jakarta
- Spain (4):
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Fundación Díaz, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo RF, Ward PA. Role of C5a in inflammatory responses. Annu Rev Immunol. 2005;23:821-52. doi: 10.1146/annurev.immunol.23.021704.115835. PMID 15771587
- [Background] Wood AJT, Vassallo A, Summers C, Chilvers ER, Conway-Morris A. C5a anaphylatoxin and its role in critical illness-induced organ dysfunction. Eur J Clin Invest. 2018 Dec;48(12):e13028. doi: 10.1111/eci.13028. Epub 2018 Oct 15. PMID 30229880
- [Background] Wang R, Xiao H, Guo R, Li Y, Shen B. The role of C5a in acute lung injury induced by highly pathogenic viral infections. Emerg Microbes Infect. 2015 May;4(5):e28. doi: 10.1038/emi.2015.28. Epub 2015 May 6. PMID 26060601
- [Background] Sun S, Zhao G, Liu C, Fan W, Zhou X, Zeng L, Guo Y, Kou Z, Yu H, Li J, Wang R, Li Y, Schneider C, Habel M, Riedemann NC, Du L, Jiang S, Guo R, Zhou Y. Treatment with anti-C5a antibody improves the outcome of H7N9 virus infection in African green monkeys. Clin Infect Dis. 2015 Feb 15;60(4):586-95. doi: 10.1093/cid/ciu887. Epub 2014 Nov 27. PMID 25433014
- [Background] Sun S, Zhao G, Liu C, Wu X, Guo Y, Yu H, Song H, Du L, Jiang S, Guo R, Tomlinson S, Zhou Y. Inhibition of complement activation alleviates acute lung injury induced by highly pathogenic avian influenza H5N1 virus infection. Am J Respir Cell Mol Biol. 2013 Aug;49(2):221-30. doi: 10.1165/rcmb.2012-0428OC. PMID 23526211
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15771587/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30229880/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26060601/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25433014/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23526211/